CLINICAL TRIAL: NCT03794336
Title: Efficacy and Safety of Alogliptin vs. Acarbose in Chinese T2DM Patients With High CV Risk or CHD Treated With Aspirin and Inadequately Controlled With Metformin Monotherapy or Drug Naive: A Multicenter, Randomized, Open Label, Prospective Study
Brief Title: Efficacy and Safety of Alogliptin vs. Acarbose in Chinese Type 2 Diabetes Mellitus (T2DM) Patients With High CV Risk or CHD Treated With Aspirin and Inadequately Controlled With Metformin Monotherapy or Drug Naive
Acronym: ACADEMIC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALOGLC08867; U1111-1210-0679 (Other: UTN)
Record Dates: First submitted 2019-01-03; First posted 2019-01-07 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — alogliptin; Acarbose; Metformin; Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Alogliptin (Experimental): Single dose of alogliptin once daily for 16 weeks
  Interventions: Drug: Alogliptin; Drug: Metformin; Drug: Aspirin
- Acarbose (Active Comparator): Thrice daily dose of acarbose Dose 1 for 7 days then titrate to thrice daily dose of of acarbose Dose 2
  Interventions: Drug: Acarbose; Drug: Metformin; Drug: Aspirin

INTERVENTIONS:
Drug: Alogliptin — Pharmaceutical form: tablet
  Route of administration: oral administration
  Other Names: Nesina
  Arms: Alogliptin
Drug: Acarbose — Pharmaceutical form: tablet
  Route of administration: oral administration
  Other Names: Glucobay
  Arms: Acarbose
Drug: Metformin — Pharmaceutical form: tablet
  Route of administration: oral administration
Drug: Aspirin — Pharmaceutical form: tablet
  Route of administration: oral administration
  Other Names: Bayaspirin

SUMMARY:
Primary Objectives:

* To assess efficacy in terms of change from baseline in Hemoglobin A1c (HbA1c) at the end of study between the two drugs.
* To assess tolerability in terms of overall Gastrointestinal (GI) tolerability for Alogliptin compared with acarbose during the whole treatment period.

Secondary Objectives:

* To assess efficacy in terms of the percentage of patients achieving HbA1c<7%.
* To assess efficacy in terms of percentage of patients achieving HbA1c<7% without GI effects.
* To assess change from baseline in Fasting plasma glucose (FPG), 2-h Post plasma glucose (2-h PPG), β-cell function (HOMA-β), lipids and body weight.
* To assess safety in terms of occurrence of hypoglycemia events.
* To assess safety in terms of other adverse events.
* To assess patient adherence and tolerability.

DETAILED DESCRIPTION:
The duration of the study for each patient will be approximately 17 weeks consisting of about 1 week screening period and 16-week treatment period.

ELIGIBILITY:
Inclusion criteria :

* Type 2 Diabetes Mellitus patients (age ≥18yr) drug naive or treated with metformin monotherapy (≥1500 mg/day or individually maximally tolerated dose) for at least 12 weeks with a Hemoglobin A1c between ≥ 7.5% and ≤ 11.0% at screening.
* Fasting plasma glucose ≤13.3mmol/L(≤240mg/dL) at screening.
* Patients with documented history of Coronary Heart Disease (CHD) or High cardiovascular(CV) risk.
* History of CHD, defined as previous myocardial infarction or unstable/stable angina.
* High CV risk, defined as male or female (age> 50 yr), combined with at least one of these risk factors as below: family history of cardiovascular disease, history of hypertension, smoking, dyslipidemia, or protein urine.
* Already treated with Aspirin or should start Aspirin treatment at physician's discretion.

Exclusion criteria:

* Diagnosis of type 1 diabetes, diabetes resulting from pancreatic injury or secondary forms of diabetes.
* Previous treatment with any Dipeptidyl Peptidase -4 inhibitor or glucagon-like peptide-1 (GLP-1) receptor agonists within 1 year of screening;
* Any contraindication of Aspirin, Dipeptidyl Peptidase- 4 inhibitor and Alpha-glucosidase inhibitor.
* Clinically apparent liver disease or moderate /severe renal impairment or end-stage renal disease
* Unstable CV disorder including heart failure (New York Heart Association class III or IV), refractory angina, uncontrolled arrhythmias, and severe uncontrolled hypertension (systolic blood pressure ≥180 mmHg, or diastolic blood pressure ≥105 mmHg).
* Acute coronary syndrome event within 6 month before randomization

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1293 (Actual)
Dates: Start 2019-06-29 (Actual); Primary Completion 2020-12-14 (Actual); Study Completion 2020-12-14 (Actual)

PRIMARY OUTCOMES:
Change in Hemoglobin A1c | Baseline to week 16
  Change from baseline in Hemoglobin A1c at the end of study (week 16) between the two drugs
Overall Gastrointestinal tolerability | Baseline to week 16
  Incidence of any gastrointestinal adverse events during the whole treatment period.

SECONDARY OUTCOMES:
Percentage of patients achieving HbA1c <7% | Baseline to Week 16
  Percentage of patients achieving HbA1c <7% at the end of study
Percentage of patients achieving HbA1c <7% without gastrointestinal effects | Baseline to Week 16
  Percentage of patients achieving HbA1c <7% without gastrointestinal effects at the end of study
Change in Fasting Plasma Glucose (FPG) | Baseline to Week 16
  Change in FPG from baseline to week 16 between the two groups of drugs
Occurrence of hypoglycemia events | Baseline to Week 16
  Number of patients reporting hypoglycemia events
Other Adverse Events (AEs) | Baseline to Week 16
  Number of patients reporting other Adverse Events
Overall tolerability | Baseline to Week 16
  Percentage of patients who discontinued study treatment as a result of adverse drug reaction
Change in Postprandial Plasma Glucose 2-h (PPG) | Baseline to Week 16
  Change in PPG from baseline to week 16 between two groups of drug
Change in Homeostasis model assessment-β (HOMA- β) | Baseline to Week 16
  Change in HOMA- β from baseline to week 16 between two groups of drug
Change in Total Cholesterol (TC) | Baseline to Week 16
  Changes from baseline in TC to week 16 between the two groups
Change in Tri Glycerides (TG) | Baseline to Week 16
  Changes from baseline in TG to week 16 between the two groups
Change in High Density Lipoprotein-Cholesterol (HDL-C) | Baseline to Week 16
  Changes from baseline in HDL-C to week 16 between the two groups
Change in Low Density Lipoprotein-Cholesterol (LDL-C) | Baseline to Week 16
  Changes from baseline in LDL-C to week 16 between the two groups.
Change in body weight | Baseline to Week 16
  Changes from baseline in body weight to week 16 between the two groups
Overall adherence to Investigational Medicinal Product (IMP) | Baseline to Week 16
  Calculated as overall dosing actually taken IMPs divided by the expected overall dosing as per protocol
Medication possession ratio (MPR) | Baseline to Week 16
  Calculated as number of days actually taken IMPs divided by the expected number of days as per protocol

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- CHINA, China, China

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Background] Gao B, Gao W, Wan H, Xu F, Zhou R, Zhang X, Ji Q. Efficacy and safety of alogliptin versus acarbose in Chinese type 2 diabetes patients with high cardiovascular risk or coronary heart disease treated with aspirin and inadequately controlled with metformin monotherapy or drug-naive: A multicentre, randomized, open-label, prospective study (ACADEMIC). Diabetes Obes Metab. 2022 Jun;24(6):991-999. doi: 10.1111/dom.14661. Epub 2022 Mar 22. PMID 35112779